CLINICAL TRIAL: NCT01268891
Title: Randomised, Double-blind, Parallel-group, Placebo-controlled, Fixed-dose Study of [Azilect®] Rasagiline in Levodopa-treated Parkinson's Patients With Motor Fluctuations in Korea
Brief Title: Study of Azilect® (Rasagiline) in Levodopa-treated Parkinson's Disease Patients With Motor Fluctuations in Korea
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: H. Lundbeck A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 13484A
Record Dates: First submitted 2010-12-30; First posted 2010-12-31 (Estimated); Results first posted 2013-12-03 (Estimated); Last update posted 2013-12-03 (Estimated); Status verified 2013-10

CONDITIONS: Parkinson's Disease
Keywords: Azilect; Motor fluctuations; Parkinson´s Disease; Rasagiline
MeSH Terms: conditions — Parkinson Disease | interventions — rasagiline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Azilect® (Experimental)
  Interventions: Drug: Azilect®

INTERVENTIONS:
Drug: Placebo — Once daily; tablet; orally; 18 weeks
  Arms: Placebo
Drug: Azilect® — 1 mg daily; tablet; orally; 18 weeks
  Other Names: Rasagiline
  Arms: Azilect®

SUMMARY:
To evaluate the efficacy of a fixed dose of Azilect® (1 mg/day) vs placebo as assessed by the change from baseline in mean total daily OFF time during 18 weeks of treatment in levodopa-treated Parkinson's Disease (PD) patients with motor fluctuations in Korea.

DETAILED DESCRIPTION:
Levodopa has been the mainstay therapy for PD for decades, and it is considered to be one of the most effective medications for relief of the symptoms of PD. However, within few months to few years the majority of levodopa-treated patients notice a decline in the duration of benefit of each dose and develop motor-complications. A major problem is the appearance of fluctuations in mobility, cycles of ON and OFF periods. The administration of Azilect®, a monoamine oxidase type B (MAO-B) inhibitor, can slow the elimination of the endogenous dopamine supplies or the dopamine produced from the exogenous levodopa therapy and may therefore improve ON-OFF fluctuations. Azilect® is approved for treatment of PD in Europe and the US.

The objective of this study is to evaluate the efficacy, tolerability, and safety of Azilect® compared to placebo in Korean PD patients with motor fluctuations on levodopa therapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients with idiopathic PD
* Patients with motor fluctuations averaging at least 1 hour daily in the OFF state during the waking hours (not including morning akinesia)
* Patients with a Modified Hoehn and Yahr stage <5 in the OFF state
* Patients taking optimised levodopa/DOPA decarboxylase inhibitor (DDI) therapy for at least 14 days prior to baseline
* Patients receiving at least 3 daily doses of levodopa, not including a bedtime dose, and not more than 8 daily doses of levodopa
* Patient who have demonstrated the ability to keep accurate 24-hour diaries prior to randomisation

Exclusion Criteria:

* Patients with a clinically significant or unstable medical or surgical condition that would preclude his/her safe and complete study participation
* Patients taking any disallowed medication according to the Azilect® approved label
* Patients taking MAO inhibitors within 3 months prior to baseline visit
* Patients with a known serious adverse reaction to selegiline
* Patients with a clinically significant psychiatric illness, including a major depression, which compromises their ability to provide consent or participate fully in the study
* Patients with a Mini Mental State Examination (MMSE) score <=24
* Patients with a diagnosis of melanoma or a history of melanoma, or a suspicious lesion

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2011-01; Primary Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Email contact via H. Lundbeck A/S, Study Director — LundbeckClinicalTrials@lundbeck.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study consisted of a 2-week Screening Period during which the levodopa dose was optimised (if required), a 2-week Screening Period during which the levodopa dose was stabilised, an 18-week double-blind treatment period with rasagiline or placebo once daily (patients were randomised in a 1:1 ratio), and a 4-week Safety Follow-up Period.
Period: Overall Study
Arm/Group | Placebo | Azilect®
Started | 66 | 66
Completed | 58 | 58
Not Completed | 8 | 8
Not completed — Adverse Event | 3 | 7
Not completed — Lack of Efficacy | 1 | 0
Not completed — Withdrawal of Consent | 3 | 1
Not completed — Administrative or other reason(s) | 1 | 0

BASELINE CHARACTERISTICS:
Population: Age and Gender: all-patients-treated set (APTS) - all patients in the APRS who took at least one dose of investigational medicinal product (IMP).
  Study-specific Characteristics: full-analysis set (FAS) - all patients in the APTS who had at least one valid post-baseline assessment of total daily OFF time (at least one valid post-baseline diary).
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Azilect® | Total
Number analyzed (Participants) | 66 | 66 | 132
Age Continuous [Mean (Standard Deviation); unit: years] | 59.5 (9.0) | 60.2 (8.6) | 59.8 (8.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 33 | 56
  Male | 43 | 33 | 76
Total Daily OFF Time [Mean (Standard Deviation); unit: hours] — Parkinson's Disease Patient Diary is a self-administered diary designed to assess motor fluctuations throughout the day. It is divided into 30-minute intervals, and the patient selects one of four options for each interval: asleep; off; on with no dyskinesia or without troublesome dyskinesia; or on with troublesome dyskinesia.
  hours | 6.24 (2.73) | 6.26 (2.29) | 6.25 (2.50)
CGI-S [Mean (Standard Deviation); unit: units on a scale] — Clinical Global Impression - Severity of Illness (CGI-S) is a single-item rating scale used to evaluate a patient's severity of illness on a 7-point scale, based on the investigator's total clinical experience with patients. The scale ranges from 1 (normal, not at all ill) to 7 (among the most extremely ill patients).
  units on a scale | 3.05 (0.92) | 2.94 (1.11) | 2.99 (1.02)
UPDRS-ADL Score During OFF Time [Mean (Standard Deviation); unit: units on a scale] — Unified Parkinson's Disease Rating Scale (UPDRS) is a 42-item rating scale designed to assess Parkinson's Disease-related disability and impairment using a patient interview and a physical examination. It has 4 parts and 4 subsection scores. A higher score indicates a worst outcome. I: mentation, behaviour and mood symptoms - 0 to 16; II: activities of daily living (ADL) - 0 to 52; III: motor function - 0 to 108; IV: complications of dopaminergic therapy - 0 to 23. Subsection scores for I to III are used to calculate a total score that ranges from 0 (no disability) to 176 (total dependence).
  units on a scale | 11.15 (5.84) | 11.79 (6.58) | 11.48 (6.21)
UPDRS Motor Score During ON time [Mean (Standard Deviation); unit: units on a scale] — UPDRS is a 42-item rating scale designed to assess Parkinson's Disease-related disability and impairment using a patient interview and a physical examination. It has 4 parts and 4 subsection scores. A higher score indicates a worst outcome. I: mentation, behaviour and mood symptoms - 0 to 16; II: ADL - 0 to 52; III: motor function - 0 to 108; IV: complications of dopaminergic therapy - 0 to 23. Subsection scores for I to III are used to calculate a total score that ranges from 0 (no disability) to 176 (total dependence).
  units on a scale | 19.81 (8.39) | 17.98 (8.71) | 18.86 (8.57)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Mean Total Daily OFF Time Using Parkinson's Disease Patient Diary
Description: Parkinson's Disease Patient Diary is a self-administered diary designed to assess motor fluctuations throughout the day. It is divided into 30-minute intervals, and the patient selects one of four options for each interval: asleep; off; on with no dyskinesia or without troublesome dyskinesia; or on with troublesome dyskinesia.
  The Change From Baseline in Mean Total Daily OFF Time is calculated by taking the difference between the average of the total daily OFF time at Weeks 6, 10, 14 and 18, and the Baseline Total Daily OFF Time.
Time Frame: Baseline and Weeks 6, 10, 14, and 18
Population: Full-analysis set (FAS); observed cases (OC)
Measure: Mean (Standard Error); unit: hours
Arm/Group | Placebo | Azilect®
Number analyzed (Participants) | 59 | 63
hours | -1.24 (0.26) | -1.59 (0.25)
Statistical Analysis 1: Comparison: Placebo vs Azilect®; The power for this study, which is designed to show a trend, that is, to show a clinical difference in the primary outcome measure, is 72%; Test type: Superiority or Other; p = 0.3257, ANCOVA — The threshold for statistical significance in showing a trend for this study is 0.10; Mean Difference (Final Values) = -0.35, 90% CI 2-sided [-0.93 to 0.23], Standard Error of Mean 0.35

2. Secondary Outcome: Clinical Status Using CGI-I Score During ON Time
Description: Clinical Global Impression - Global Improvement (CGI-I) is a single-item rating scale used to evaluate a patient's condition relative to baseline on a 7-point scale, regardless of whether the improvement is related to the investigational medicinal product (IMP). The scale ranges from 1 (very much improved) to 7 (very much worse).
Time Frame: Week 18
Population: FAS; last observation carried forward (LOCF)
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Azilect®
Number analyzed (Participants) | 59 | 63
units on a scale | 3.35 (0.13) | 3.05 (0.13)
Statistical Analysis 1: Comparison: Placebo vs Azilect®; Test type: Superiority or Other; p = 0.0946, ANCOVA; Mean Difference (Final Values) = -0.30, 95% CI 2-sided [-0.65 to 0.05], Standard Error of Mean 0.18

3. Secondary Outcome: Change From Baseline in UPDRS-ADL Score During OFF Time
Description: Unified Parkinson's Disease Rating Scale (UPDRS) is a 42-item rating scale designed to assess Parkinson's Disease-related disability and impairment using a patient interview and a physical examination. It has 4 parts and 4 subsection scores. A higher score indicates a worst outcome. I: mentation, behaviour and mood symptoms - 0 to 16; II: activities of daily living (ADL) - 0 to 52; III: motor function - 0 to 108; IV: complications of dopaminergic therapy - 0 to 23. Subsection scores for I to III are used to calculate a total score that ranges from 0 (no disability) to 176 (total dependence).
Time Frame: Baseline and Week 18
Population: FAS; LOCF
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Azilect®
Number analyzed (Participants) | 59 | 63
units on a scale | 0.13 (0.42) | -0.57 (0.41)
Statistical Analysis 1: Comparison: Placebo vs Azilect®; Test type: Superiority or Other; p = 0.2258, ANCOVA; Mean Difference (Final Values) = -0.70, 95% CI 2-sided [-1.84 to 0.44], Standard Error of Mean 0.57

4. Secondary Outcome: Change From Baseline in UPDRS Motor Score During ON Time
Description: UPDRS is a 42-item rating scale designed to assess Parkinson's Disease-related disability and impairment using a patient interview and a physical examination. It has 4 parts and 4 subsection scores. A higher score indicates a worst outcome. I: mentation, behaviour and mood symptoms - 0 to 16; II: ADL - 0 to 52; III: motor function - 0 to 108; IV: complications of dopaminergic therapy - 0 to 23. Subsection scores for I to III are used to calculate a total score that ranges from 0 (no disability) to 176 (total dependence).
Time Frame: Baseline and Week 18
Population: FAS; LOCF
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Azilect®
Number analyzed (Participants) | 59 | 63
units on a scale | -1.52 (0.72) | -2.87 (0.69)
Statistical Analysis 1: Comparison: Placebo vs Azilect®; Test type: Superiority or Other; p = 0.1700, ANCOVA; Mean Difference (Final Values) = -1.35, 95% CI 2-sided [-3.29 to 0.59], Standard Error of Mean 0.98

ADVERSE EVENTS:
Time Frame: Serious Adverse Events: 18-week double-blind treatment period and 4-week safety follow-up period. Other Adverse Events: 18-week double-blind treatment period.
Arm/Group | Placebo | Azilect®
Serious Adverse Events (participants affected / at risk) | 4/66 | 5/66
Other Adverse Events (participants affected / at risk) | 12/66 | 19/66
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Placebo (N=66) | Azilect® (N=66)
Gastritis (Gastrointestinal disorders) | 0 | 1
Pyelonephritis acute (Infections and infestations) | 0 | 1
Joint injury (Injury, poisoning and procedural complications) | 1 | 0
Subdural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Wrist fracture (Injury, poisoning and procedural complications) | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Borderline ovarian tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/23 | 1/33
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Loss of consciousness (Nervous system disorders) | 0 | 1
Subarachnoid haemorrhage (Nervous system disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=66) | Azilect® (N=66)
Accidental overdose (Injury, poisoning and procedural complications) | 5 | 3
Dizziness (Nervous system disorders) | 1 | 4
Dyskinesia (Nervous system disorders) | 5 | 8
Insomnia (Psychiatric disorders) | 2 | 4
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The results of this study will be published at the discretion of H. Lundbeck A/S. H. Lundbeck A/S will ensure that the authorship of all publications based on this study is in accordance with the criteria defined by the International Committee of Medical Journal Editors (ICMJE).

The primary publication must be published before any secondary publications.